CLINICAL TRIAL: NCT06588803
Title: A Long-term Follow-up Study Evaluating Intravenous Injection of EXG001-307 in Patients With Type 1 Spinal Muscular Atrophy (SMA)
Brief Title: A Long-term Follow-up Study Evaluating Intravenous Injection of EXG001-307 in Patients With Type 1 SMA
Status: Enrolling by invitation | Type: Observational
Sponsor: Hangzhou Jiayin Biotech Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: EXG001-307-LTFU
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: SMA
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Single Person

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, only for observational studies — No intervention, only for observational studies

SUMMARY:
An Open-label, Long-term Follow-Up Study to Evaluate the Safety and Tolerability of Gene Therapy with EXG001-307 in SMA1 patients ,who joined the parent study (EXG001-307-102)

DETAILED DESCRIPTION:
This study plans to enroll type 1 SMA patients who have previously received EXG001-307 treatment in the parent trial EXG001-307-102 to observe the long-term safety and efficacy of gene therapy with EXG001-302.

The first year of long-term follow-up will be conducted every 3 months ; In the second year, follow-up visits will be conducted every six months, with telephone follow ups at 15 and 21 months during this period; From 3 to 5 years after gene therapy, follow up by phone every six months and follow on on site once a year.

ELIGIBILITY:
Inclusion Criteria:

1. Previously received treatment with EXG001-307 in trial EXG001-307-102;
2. Parents or guardians understand the research procedure and sign the ICF; Good compliance and willingness to follow research procedures. Voluntarily participate in this clinical trial.

Exclusion Criteria:

1. Parents or guardians are unwilling or unable to participate in long-term follow-up studies.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 1 SMA patients who have previously used EXG001-307 in trial EXG001-307-102 .
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2030-09-10 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
long-term safety：Assess the types, severity, and incidence of serious adverse events (SAEs) and adverse events of particular concern (AESIs) | 4 years
  Assess the types, severity, and incidence of serious adverse events (SAEs) and adverse events of particular concern (AESIs)

SECONDARY OUTCOMES:
Evaluate the long-term effectiveness of EXG001-307 treatment: assess the achievement of exercise milestones based on the scale | 4 years
  The achievement of new milestones in the third edition of the Berry Infant and Child Development Scale (BSID-III)：
  Doctors need to evaluate whether patients can achieve the following milestones:
  head control：Can children keep their heads upright for at least 3 seconds without support； sitting without assistant：Can children sit up alone for at least 5 seconds without support； standing with assistant：Can children use chairs or other convenient objects as support to stand up on their own； standing without assistant：Can the child stand alone for at least 3 seconds after the evaluator releases the child's hand； walking with assistant：Can children make coordinated and alternating stepping movements while walking； walking without assistant：Can children walk at least three steps without support, even if their gait is stiff and unstable；
Evaluate the long-term effectiveness of EXG001-307 treatment: evaluate event free survival rate | 4 years
  Event free survival rate:
  The event free survival rate refers to the proportion of subjects who did not die and did not require permanent mechanical ventilation with a ventilator. Permanent mechanical ventilation refers to the need for tracheotomy to maintain ventilation in irreversible emergencies or after emergency resolution, or the need to rely on Bipap mechanical ventilation support for ≥ 16 hours per day for more than 3 consecutive weeks, or tracheal intubation for ≥ 3 weeks; Researchers evaluate patients by examining their daily use of ventilators.
Evaluate the immunogenicity of EXG001-307 after treatment, including measuring the titers of anti-AAV9-ADA and anti-SMN-ADA antibodies. | 4 years
  After blood collection, send it to the central laboratory to complete the following antibody testing: the titers of anti-AAV9-ADA and anti-SMN-ADA antibodies (until two consecutive negative results);
Evaluate the distribution of viral vectors after treatment with EXG001-307: detect the level of vector genome in saliva, feces, and urine samples of subjects. | 4 years
  Carrier distribution: Genomic level of carriers in saliva, urine, and fecal samples (up to two consecutive negative resultst);
Exploratory objective: To calculate the proportion of subjects receiving other SMA treatments during the trial period | 4 years
  Calculate the proportion of subjects receiving other SMA treatments to the total number of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: YI WANG, Ph D., Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- The Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No